CLINICAL TRIAL: NCT04693273
Title: Novel Decision Aid for Carpal Tunnel Patients: Exploring Patient Preferences Between WALANT and Traditional Surgery
Brief Title: Novel Decision Aid for Carpal Tunnel Patients
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Charles S Day, Professor & Executive Vice Chair of the Orthopaedic Service Line, Henry Ford Health System
Other Study IDs: 13583
Record Dates: First submitted 2020-12-16; First posted 2021-01-05 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: WALANT; Wide-Awake-Local-Anesthesia-no-Tourniquet
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Decision Support Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carpal Tunnel Release surgical patients: This is the group the investigators survey who are candidates for carpal tunnel release (CTR) surgery: patients should be 18 years or older, comprehend and read English, and patients who consent to do the survey.
  Interventions: Other: Decision Aid for Surgical Modality Choice

INTERVENTIONS:
Other: Decision Aid for Surgical Modality Choice — A novel decision aid that helps surgical patients choose between Wide-Awake carpal tunnel release and traditional tourniquet surgery. It involves an orientation-memory-concentration test to test if patients are cognitively capable of making decisions, then the decision aid table that has similarities and differences between the two modalities, and a few survey questions that help the investigators know what the patients prefer. Finally, patients finish the decision conflict test to see how confident these patients are about their preference.

SUMMARY:
A questionnaire will be given to patients who are considering undergoing hand surgery as a treatment for Carpal Tunnel Syndrome to help participants decide between two surgical options- Wide-Awake-Local-Anesthesia-no-Tourniquet (WALANT) and traditional open hand surgery. These patients will be asked to complete a pre-questionnaire knowledge test and a post-questionnaire knowledge test. the primary objective is to validate this questionnaire to be used by other orthopedic surgeons. This study will also reveal patient preference between these two surgical treatments for carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of older,
* CTS patients who are CTR candidates,
* Comprehend and understand English,
* Passed the Orientation-memory-concentration test done before the decision aid

Exclusion Criteria:

* Younger than 18 years of age,
* Non-CTS patients,
* Not CTR candidates,
* Do not comprehend or read English,
* Failed the Orientation-memory-concentration test done before the decision aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are CTR candidates will be asked to participate in this study considering such patients are 18 years or older, comprehend and read English, and considering the participation depends on passing the orientation, concentration, and memory test.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Surgical Modality preference for CTR through questionnaire answers | Feb, 2020- Feb, 2021
  Investigators will reveal participants' preferences regarding the preferred surgical modality between WALANT and traditional tourniquet by having a questionnaire question after participants read the decision aid whereby such participants are asked whether their preference is WALANT or traditional tourniquet carpal tunnel release after having learned about both.

SECONDARY OUTCOMES:
Patient Knowledge scores Before the decision aid use | Feb, 2020- Feb, 2021
  This is achieved through 4 multiple-choice questions (the score is out of 4) that are completed by the patient before reading the decision aid. The questions revolve around concepts relevant to wide-awake and traditional-tourniquet carpal tunnel release surgical modalities. These questions assess the patient's prior knowledge.
Patient knowledge scores after the decision aid use | Feb, 2020- Feb, 2021
  This is achieved through 4 multiple-choice questions (the score is out of 4) that are completed by the patient after reading the decision aid. They are the same questions as those done before the decision aid but aim to test if the patient truly understood and learned from the decision tool. This knowledge score along with the score of the questions done before the decision aid will help assess if a significant enhancement of the knowledge scores happened which reflects a useful decision aid.
Decisional Conflict Score | Feb, 2020- Feb, 2021
  A previously validated scale was used which involves several questions assessing how confident the patient is about the decision/preference declared and how much it resembles their values. Patients are asked to assess their agreement/disagreement on several factors on the scale using a Likert scale between 0 (confident) and 4 (not confident ). The lower the aggregate score, the more confident the participant is. Per the scale's manual, a score of 25 or lower reflects a confident patient while any score over 36 reflects decisional hesitation or conflict. (This is the reference for the decisional scale's manual that is used in the study: https://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decisional_Conflict.pdf)

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Day, M.D., M.B.A., Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Patient information will be de-identified and then will be deleted after completion of the study. Patient information will not be shared with others.